CLINICAL TRIAL: NCT07237802
Title: Efficacy of an Online Pain Neuroscience Education Intervention in Women With Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Online Pain Neuroscience Education for Women With Primary Dysmenorrhea
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Dr, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIVERSITYCARDENALHERRERA-100
Record Dates: First submitted 2025-10-01; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Primary Dysmenorrhea (PD)
Keywords: Pain; Dysmenorrhea; Kinesiophobia
MeSH Terms: conditions — Pain; Dysmenorrhea; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Individually randomized, two-arm parallel trial (1:1) comparing an online pain neuroscience education (PNE) program plus lifestyle recommendations with lifestyle recommendations alone in women with primary dysmenorrhea. Randomization will be computer-generated and allocation concealed by an independent researcher. Outcomes will be assessed at baseline and at 6-month follow-up by blinded assessors/analysts. Intention-to-treat analysis will be applied.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors and data analysts will be blinded to group allocation. Participants and intervention providers will not be masked due to the nature of the educational program. Allocation will be concealed using a computer-generated randomization sequence managed by an independent researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Pain Neuroscience Education (PNE) (Experimental): Participants in this arm will receive an online pain neuroscience education (PNE) program plus usual lifestyle recommendations. The PNE intervention consists of four weekly audiovisual and written modules adapted to the context of primary dysmenorrhea, focusing on the neurobiology and biopsychosocial aspects of pain, with practical strategies to reduce maladaptive beliefs, kinesiophobia, and catastrophizing.
  Interventions: Other: PNE online + lifestyle recommendations.
- Active Comparator (Active Comparator): Participants in this arm will receive the usual lifestyle recommendations for primary dysmenorrhea. These recommendations include general advice on healthy habits and self-management strategies typically provided in clinical practice.
  Interventions: Other: Lifestyle recommendations

INTERVENTIONS:
Other: PNE online + lifestyle recommendations. — Four-week online educational program with audiovisual modules on the neurobiology and biopsychosocial aspects of pain, adapted to women with primary dysmenorrhea. In addition, participants receive usual lifestyle recommendations, including general advice on healthy habits and self-management strategies commonly provided in clinical practice.
  Arms: Online Pain Neuroscience Education (PNE)
Other: Lifestyle recommendations — Participants in this arm will receive online lifestyle recommendations for four weeks, including general advice on healthy habits and self-management strategies commonly provided in clinical practice for women with primary dysmenorrhea.
  Arms: Active Comparator

SUMMARY:
Primary dysmenorrhea is a highly prevalent condition characterized by recurrent menstrual pain in the absence of identifiable pelvic pathology. It affects up to 95% of menstruating women and often interferes with quality of life. Pain neuroscience education (PNE) has shown positive effects in musculoskeletal conditions but has not yet been studied in women with primary dysmenorrhea. This study aims to evaluate the effect of an online PNE intervention combined with lifestyle recommendations, compared to lifestyle recommendations alone

DETAILED DESCRIPTION:
This randomized controlled trial will compare an online pain neuroscience education (PNE) program plus lifestyle recommendations with lifestyle recommendations alone in women with primary dysmenorrhea. Participants will be randomized (1:1) to either the intervention group (4-week online PNE modules plus lifestyle recommendations) or the control group (lifestyle recommendations only). The program is based on Butler and Moseley's pain neuroscience principles, adapted to menstrual pain. Outcomes will be assessed at baseline and at 6 months. The primary outcome is pain intensity. Secondary outcomes include anxiety, depression, kinesiophobia and pain catastrophizing,

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women aged 18 to 35 years.
* Clinical diagnosis of primary dysmenorrhea.
* History of moderate to severe menstrual pain for at least six consecutive menstrual cycles.
* Pain intensity score greater than 5 on a numerical rating scale (0-10).
* No prior use of pain neuroscience education (PNE).
* No history of pregnancy.

Exclusion Criteria:

* History of lower abdominal surgery.
* Presence of severe mental health disorders.
* Current use of hormonal contraceptives.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured by the 11-point Numeric Rating Scale (NRS) | pre-intervention and 6 months post-intervention
  Pain intensity will be assessed using the 11-point Numeric Rating Scale (NRS). Participants will rate their average menstrual pain intensity over the previous cycle, from 0 ("no pain") to 10 ("worst imaginable pain"). Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Anxiety and depression measured by the Hospital Anxiety and Depression Scale (HADS) | pre-intervention and 6 months post-intervention
  The Hospital Anxiety and Depression Scale (HADS) has 14 items, with two subscales: HADS-Anxiety (7 items) and HADS-Depression (7 items). Each subscale ranges 0-21; higher scores indicate greater anxiety/depression.
Kinesiophobia measured by the Tampa Scale for Kinesiophobia-11 (TSK-11) | pre-intervention and 6 months post-intervention
  The Tampa Scale for Kinesiophobia-11 (TSK-11) has 11 items scored 1 ("strongly disagree") to 4 ("strongly agree"). Total score 11-44; higher scores indicate greater fear of movement/re-injury.
Pain catastrophizing measured by the Pain Catastrophizing Scale (PCS) | pre-intervention and 6 months post-intervention
  The Pain Catastrophizing Scale (PCS) includes 13 items scored 0 ("not at all") to 4 ("all the time"). Total score 0-52; higher scores indicate greater pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Lisón Párraga, Dr, Principal Investigator — Universidad Cardenal Herrera CEU
Locations (1):
- Universidad CEU Cardenal Herrera, Valencia, Valencia-valència, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Soderman L, Edlund M, Marions L. Prevalence and impact of dysmenorrhea in Swedish adolescents. Acta Obstet Gynecol Scand. 2019 Feb;98(2):215-221. doi: 10.1111/aogs.13480. Epub 2018 Nov 6. PMID 30312470
- [Background] Butler DS, Moseley GL. Explain Pain. 2nd ed. Adelaide, South Australia: Noigroup Publications; 2013.